CLINICAL TRIAL: NCT02449538
Title: Study to Evaluate the Safety and Efficacy of Everolimus, in Subjects With PIK3CA Amplification, PTEN Loss and PIK3CA Mutation Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01-117
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- everolimus (Experimental): everolimus 10 mg qd daily
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — everolimus 10 mg qd daily one cycle is 28days.
  Other Names: RAD001

SUMMARY:
This study is a single-arm, phase II study of everolimus in patients with PTEN loss ,PIK3CA mutation and PIK3CA amplification Refractory Solid Tumors .

Everolimus 10 mg will be administered orally qd daily.

To investigate the efficacy and safety of everolimus in patients with PTEN loss ,PIK3CA mutantion and PIK3CA amplification Refractory Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. PIK3CA amplification, PTEN loss and PIK3CA mutation Refractory Solid Tumors that has recurred or progressed following standard therapy, or that has not responded to standard therapy, or for which there is no standard therapy.
4. ECOG performance status 0-2.
5. Have measurable or evaluated disease based on RECIST1.1. as determined by investigator.
6. Adequate Organ Function Laboratory Values

   * Absolute neutrophil count ≥ 1.5 x 109/L, Hemoglobin ≥ 9g/dL, Platelets ≥ 75 x 109/L
   * bilirubin ≤ 1.5 x upper limit of normal AST/ALT ≤ 2.5 x upper limit of normal (5.0 X upper limit of normal , for subjects with liver metastases)
   * creatinine ≤1.5 x UNL
7. Patients of child-bearing potential should be using adequate contraceptive measures (two forms of highly reliable methods) should not be breast feeding and must have a negative pregnancy test prior to start of dosing.
8. Adequate heart function.

Exclusion Criteria:

1. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
2. Has known active central nervous system (CNS) metastases.
3. Has an active infection requiring systemic therapy.
4. Pregnancy or breast feeding
5. Patients with cardiac problem.
6. KRAS mutation (codon 12 or 13) or BRAF mutation (V600)
7. Any previous treatment with everolimus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
overall response rate | 24 weeks

SECONDARY OUTCOMES:
progression free survival | 24 weeks
overall survival | 24 weeks
Number of subjects with Adverse Events as a measure of toxicity profile | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jee yun Lee, MD,Ph.D., Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Samsung Medical center, Seoul, South Korea

REFERENCES:
- [Derived] Kim ST, Lee J, Park SH, Park JO, Park YS, Kang WK, Lim HY. Prospective phase II trial of everolimus in PIK3CA amplification/mutation and/or PTEN loss patients with advanced solid tumors refractory to standard therapy. BMC Cancer. 2017 Mar 23;17(1):211. doi: 10.1186/s12885-017-3196-6. PMID 28330462